CLINICAL TRIAL: NCT05497128
Title: Standard Cut Rate 27-Gauge System Versus Ultrahigh-Speed 27-Gauge System in Macular Surgery : A Randomized Controlled Trial
Brief Title: Standard Cut Rate 27-Gauge System Versus Ultrahigh-Speed 27-Gauge System in Macular Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Kyu Hyung Park, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-2112-728-001
Record Dates: First submitted 2022-08-07; First posted 2022-08-11 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Macular Disease
Keywords: Macular disease; Vitrectomy
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrahigh-speed cut rate 27-gauge system (Experimental): Patients will receive the pars plana vitrectomy in the macular disease with the 27-gauge vitrectomy systems with 20,000 cpm probes.
  Interventions: Device: Ultrahigh-speed cut rate 27-gauge system
- Standard cut rate 27-gauge system (Active Comparator): Patients will receive the pars plana vitrectomy in the macular disease with the 27-gauge vitrectomy systems with 10,000 cpm probes.
  Interventions: Device: Standard cut rate 27-gauge system

INTERVENTIONS:
Device: Ultrahigh-speed cut rate 27-gauge system — The ultrahigh-speed cut rate 27-gauge system (27+®GA HYPERVIT® Vitrectomy Probe (Alcon Laboratories, Fort Worth, TX, USA))
  Arms: Ultrahigh-speed cut rate 27-gauge system
Device: Standard cut rate 27-gauge system — The current standard cut rate 27-gauge vitrectomy system (27+®GA Advanced ULTRAVIT® Vitrectomy Probe (Alcon Laboratories, Fort Worth, TX, USA))
  Arms: Standard cut rate 27-gauge system

SUMMARY:
The purpose of this study is to compare the efficiency and safety of ultrahigh-speed cut rate 27-gauge system (27+®GA HYPERVIT® Vitrectomy Probe (Alcon Laboratories, Fort Worth, TX, USA)) and standard cut rate 27-gauge vitrectomy system (27+®GA Advanced ULTRAVIT® Vitrectomy Probe (Alcon Laboratories, Fort Worth, TX, USA)).

DETAILED DESCRIPTION:
During the last few decades, there have been dramatic changes in vitreoretinal surgery field with improvements in the performance of surgical retina equipment. As the innovation trend has been moving toward the smaller instrument calibers, the 27-gauge vitrectomy system has been developed. However, the vitrectomy system with the smaller calibers have limitations such as reduced instrument rigidity, limited availability of instrumentation, and decreased flow rate. To overcome these limitations, active developments have been ongoing to increase vitreous cutting speed, enlargement of the cutting port size, and enlargement of inner shaft to enable higher flow rates. Especially, the ultrahigh-speed cutter with improved cutting speed has the advantage of enabling safer vitrectomy because the faster cutting speed reduces retinal movement and minimizes the risk of iatrogenic retinal breaks. However, ultrahigh-speed cutting has a limitation in that it can reduce the flow rate through the vitreous cutter as it affects the duty cycle (percentage of time the cutter port is open relative to the complete cutting cycle). Therefore, the duty cycle of ultrahigh-speed cutter has also been improved so as not to delay the time for vitrectomy.

The investigators would like to evaluate the efficiency and safety of vitrectomy using a recently released ultra high-speed cut rate 27-gauge system (27+®GA HYPERVIT® Vitrectomy Probe (Alcon Laboratories, Fort Worth, TX, USA)) and a standard cut rate 27-gauge system (27+®GA Advanced ULTRAVIT® Vitrectomy Probe (Alcon Laboratories, Fort Worth, TX, USA)) by comparing the duration of vitrectomy and the rate of complications.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive eyes requiring macular surgery (i.e. epiretinal membrane, vitreomacular traction etc.) that underwent 27-gauge vitrectomy at Seoul National University Bundang Hospital (SNUBH) from September 2022 to August 2023. Patients will be randomized to receive 27-gauge vitrectomy with 20,000 cpm probes (20K group) or 27-gauge vitrectomy with 10,000 cpm probes (standard group).

Exclusion Criteria:

1. Previously vitrectomized eye
2. Trauma cases
3. Proliferative diabetic retinopathy with fibrovascular membranes
4. Retinal detachment with proliferative vitreoretinopathy
5. Macular hole
6. Endophthalmitis
7. Inability to consent for procedure

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Efficiency of core vitrectomy | During the vitrectomy
  Time to completion of core vitrectomy

SECONDARY OUTCOMES:
Intraoperative complications | During the vitrectomy
  i.e. iatrogenic retinal breaks, intraocular bleeding, retinal detachment, etc.
Postoperative complications | Postoperative period within 4 months after the vitrectomy
  i.e. intraocular bleeding, retinal detachment, etc.
Efficiency of peripheral vitrectomy | During the vitrectomy
  Time to completion of peripheral vitrectomy
Efficiency of surgery | During the surgery
  Time to completion of the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kyu Hyung Park, M.D., Ph.D., Principal Investigator — Seoul National University Bundang Hospital, Seongnam, Gyunggi-do, South Korea
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, Gyunggi-do, South Korea

REFERENCES:
- [Background] Reibaldi M, Rizzo S, Avitabile T, Longo A, Toro MD, Viti F, Saitta A, Giovannini A, Mariotti C. Iatrogenic retinal breaks in 25-gauge vitrectomy under air compared with the standard 25-gauge system for macular diseases. Retina. 2014 Aug;34(8):1617-22. doi: 10.1097/IAE.0000000000000112. PMID 24651259
- [Background] Dugel PU, Abulon DJ, Dimalanta R. Comparison of attraction capabilities associated with high-speed, dual-pneumatic vitrectomy probes. Retina. 2015 May;35(5):915-20. doi: 10.1097/IAE.0000000000000411. PMID 25621945
- [Background] Mariotti C, Nicolai M, Saitta A, Orsini E, Viti F, Skrami E, Gesuita R, Reibaldi M, Giovannini A. STANDARD CUT RATE 25-GAUGE VITRECTOMY VERSUS ULTRAHIGH-SPEED 25-GAUGE SYSTEM IN CORE VITRECTOMY: A Randomized Clinical Trial. Retina. 2016 Jul;36(7):1271-4. doi: 10.1097/IAE.0000000000000924. PMID 26702843